CLINICAL TRIAL: NCT00054028
Title: A Phase I/II Study of Suramin in Combination With Paclitaxel in Advanced (Stage IIIB or IV) Metastatic Breast Cancer
Brief Title: Suramin and Paclitaxel in Treating Women With Stage IIIB-IV Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01431; 0216; OSU-02H0216; OSU-0216; NCI-5851; CDR0000269707; U01CA076576 (NIH)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Recurrent Breast Cancer; Stage IIIB Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Suramin; Paclitaxel; Taxes

ARMS (1):
- Treatment (suramin and paclitaxel) (Experimental): PHASE I: Patients receive low-dose suramin IV over 30 minutes and paclitaxel IV over 1 hour once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive adjusted doses of suramin until a target dose is determined. The suramin target dose is defined as the dose at which at least 5 of 6 patients achieve the target plasma concentration of 10-50 uM over the duration when paclitaxel levels are therapeutic.
  PHASE II: Patients receive paclitaxel in combination with the target dose of suramin as above.
  Interventions: Drug: suramin; Drug: paclitaxel; Other: pharmacological study

INTERVENTIONS:
Drug: suramin — Given IV
  Other Names: 309 F; Antrypol; Bayer 205; Fourneau 309; Germanin
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I/II trial studies the best dose of suramin when given together with paclitaxel in treating women with stage IIIB-IV breast cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Suramin may increase the effectiveness of paclitaxel by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose of suramin in combination with paclitaxel (TXT) that results in suramin plasma concentrations approaching 10-50 uM over the duration, when TXT in the plasma is at therapeutically significant levels, in women with stage IIIB or IV breast cancer. (Phase I) II. Determine the objective response rate in patients treated with this regimen. (Phase II)

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of low-dose suramin in these patients. (Phase I) II. Determine the time to tumor progression in patients treated with this regimen. (Phase II) III. Determine the 1-year survival of patients treated with this regimen. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of suramin followed by a phase II multicenter study.

PHASE I: Patients receive low-dose suramin intravenously (IV) over 30 minutes and paclitaxel IV over 1 hour once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive adjusted doses of suramin until a target dose is determined. The suramin target dose is defined as the dose at which at least 5 of 6 patients achieve the target plasma concentration of 10-50 uM over the duration when paclitaxel levels are therapeutic.

PHASE II: Patients receive paclitaxel in combination with the target dose of suramin as above.

PROJECTED ACCRUAL: A total of 6-18 patients will be accrued for the phase I study within 9 months. A total of 28 patients will be accrued for the phase II study within 18-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IIIB or IV metastatic breast cancer (MBC)
* Prior chemotherapy:

  * Phase I: patients must have received prior paclitaxel or other taxanes in either the adjuvant or metastatic setting; prior chemotherapy, radiation or surgery must be completed at least 21 days before study entry; prior treatment with anthracyclines is not required
  * Phase II: up to two prior chemotherapy regimens for stage IIIB or IV MBC; patients must have received prior paclitaxel or other taxanes in either the adjuvant or metastatic setting; prior chemotherapy, radiation or surgery must be completed at least 21 days before study entry; prior treatment with anthracyclines is not required
* Measurable disease (phase II)
* No known brain metastases
* Hormone receptor status:

  * Not specified
* Performance status - Eastern Cooperative Oncology Group (ECOG) 0-2
* White blood cell (WBC) at least 3,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* Bilirubin no greater than 1.5 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) no greater than 2.5 times upper limit of normal
* Creatinine no greater than 1.5 mg/dL
* Left ventricular ejection fraction (LVEF) at least lower limit of normal
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributable to compounds of similar chemical or biological composition to Cremophor
* No concurrent uncontrolled illness that would preclude study compliance
* No ongoing or active infection
* No uncontrolled diabetes mellitus
* No psychiatric illness or social situations that would preclude study compliance
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No more than 2 prior chemotherapy regimens for this malignancy (phase II)
* No concurrent steroids or hormones except the following:

  * Steroids to prevent hypersensitivity reactions prior to paclitaxel administration
  * Hormones for nondisease-related conditions (e.g., insulin for diabetes)
* At least 3 weeks since prior radiotherapy and recovered
* At least 3 weeks since prior surgery and recovered
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients
* No other concurrent investigational agents
* Concurrent bisphosphonates (i.e., pamidronate or zoledronate) are allowed for the treatment of hypercalcemia or palliation of skeletal metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Shapiro, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I trial was performed at Ohio State University(OSU). Phase II, OSU was the coordinating center with other participating centers.
Pre-assignment Details: Women with metastatic breast cancer
Period: Overall Study
Arm/Group | Treatment (Suramin and Paclitaxel)
Started | 31
Phase I | 9
Phase II | 22
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Suramin and Paclitaxel (Phase I): Patients receive low-dose suramin IV over 30 minutes and paclitaxel IV over 1 hour once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive adjusted doses of suramin until a target dose is determined. The suramin target dose is defined as the dose at which at least 5 of 6 patients achieve the target plasma concentration of 10-50 uM over the duration when paclitaxel levels are therapeutic.
- Suramin and Paclitaxel (Phase II): Patients receive paclitaxel in combination with the target dose of suramin.
- Total: Total of all reporting groups
Arm/Group | Suramin and Paclitaxel (Phase I) | Suramin and Paclitaxel (Phase II) | Total
Number analyzed (Participants) | 9 | 22 | 31
Age, Continuous [Median (Full Range); unit: years] | 56 [44 to 73] | 56 [35 to 70] | 56 [35 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 22 | 31
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 8 | 19 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: patients]
  United States | 9 | 22 | 31
ECOG performance status (PS) [Number; unit: patients] — 0=Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  patients
    ECOG PS 0 | 5 | 11 | 16
    ECOG PS 1 | 4 | 8 | 12
    ECOG PS 2 | 0 | 3 | 3
Menopausal status [Number; unit: patients]
  Premenopausal | 0 | 1 | 1
  Postmenopausal | 9 | 21 | 30
ER/PR/HER 2 neu status [Number; unit: patients]
  ER+ or PR+ Status | 6 | 14 | 20
  HER2 neu+ Status | 0 | 0 | 0
  Triple negative Status | 3 | 8 | 11
Number of sites of metastastic [Number; unit: patients]
  1 | 1 | 9 | 10
  2 | 5 | 7 | 12
  ≥3 | 3 | 6 | 9
Sites of metastases [Number; unit: patients]
  Liver | 3 | 12 | 15
  Lung | 6 | 10 | 16
  Bone | 6 | 11 | 17
Prior taxane therapy [Number; unit: patients]
  Paclitaxel | 4 | 9 | 13
  Docetaxel | 5 | 10 | 15
  Nab-paclitaxel | 0 | 1 | 1
  Paclitaxel and docetaxel | 0 | 2 | 2
Prior chemotherapy (metastatic setting) [Number; unit: patients]
  0 Prior chemo therapies | 5 | 0 | 5
  1 Prior chemo therapies | 10 | 4 | 14
  2 Prior chemo therapies | 7 | 3 | 10
  3 Prior chemo therapies | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Achieved Target Suramin Concentrations in Plasma
Description: Target suramin concentration was considered achieved, if at least 5 of 6 patients achieved the target plasma concentration of 10-50 µM over the duration of 8-48 hours when paclitaxel levels are therapeutic.
Time Frame: Up to 5 years
Measure: Number; unit: percent of patients
Groups:
- Suramin and Paclitaxel: Suramin will be infused weekly over 30 minutes. Four hours after the completion of the suramin infusion the 1 hour infusion of paclitaxel will begin.
Arm/Group | Suramin and Paclitaxel
Number analyzed (Participants) | 9
percent of patients | 88

2. Primary Outcome: Objective Response Rate (Complete Response and Partial Response) as Measured by RECIST Criteria (Phase II)
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.0) for target lesion s and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR+PR.
Time Frame: Up to 8 weeks
Measure: Number; unit: patients
Arm/Group | Suramin and Paclitaxel
Number analyzed (Participants) | 22
patients
  Complete Response (CR) | 0
  Partial Response (PR) | 5

3. Secondary Outcome: Response as Measured by RECIST Criteria
Description: Evaluation of secondary endpoints will be primarily descriptive. Descriptive data will be computed and compared using analysis of variance and non-parametric rank equivalents for continuous data and chi-square or Fisher's exact test for discrete data. Response rates will include 95% confidence limits.
Time Frame: Up to 5 years
Population: Objective Response Rate
Measure: Number; unit: percentage of patients
Groups:
- Treatment (Suramin and Paclitaxel): PHASE II: Patients receive paclitaxel in combination with the target dose of suramin the same as Phase I.
Arm/Group | Treatment (Suramin and Paclitaxel)
Number analyzed (Participants) | 22
percentage of patients | 23

ADVERSE EVENTS:
Time Frame: All patients will be evaluable for toxicity using the NCI Common Toxicity Criteria version 3.0 from the time of their first treatment until the end of treatment.
Description: The NCI Common Toxicity Criteria will be used to grade and quantify toxicity events associated with therapy.
Arm/Group | Suramin and Paclitaxel
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suramin and Paclitaxel (N=31)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suramin and Paclitaxel (N=31)
Anemia (Blood and lymphatic system disorders) | 17 (17)
Anorexia (Metabolism and nutrition disorders) | 15 (15)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 15 (15)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 30 (30)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 12 (12)
Leukocytes (total WBC) (Investigations) | 14 (14)
Lymphopenia (Investigations) | 11 (11)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 14 (14)
Nausea (Gastrointestinal disorders) | 17 (17)
Neuropathy - motor (Nervous system disorders) | 5 (5)
Neuropathy-sensory (Nervous system disorders) | 26 (26)
Neutropenia (Investigations) | 8 (8)
Non-neutropenic fever (Immune system disorders) | 7 (7)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16 (16)
Renal insufficiency (Endocrine disorders) | 5 (5)
Thrombocytopenia (Injury, poisoning and procedural complications) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less